CLINICAL TRIAL: NCT03336827
Title: Improving Emotion Regulation at the End of Breast Cancer Treatment: A Randomized Controlled Study Assessing the Impact of a Multi-Component Psychological Group Intervention
Brief Title: Improving Emotion Regulation at the End of Breast Cancer Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Libre de Bruxelles (Other)
Collaborators: Jules Bordet Institute (Other); Centre de Psycho-Oncologie (CPO) (Other)
Responsible Party: Principal Investigator, Prof. Isabelle Merckaert, PhD, Professor, Université Libre de Bruxelles
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: Emotion Regulation
Record Dates: First submitted 2017-08-04; First posted 2017-11-08 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Breast Cancer; Emotional Disturbances; Emotional Dysfunction; Anxiety Depression; Fear of Cancer
Keywords: Emotion Regulation; Post-Treatment Breast Cancer Care; Cognitive-Behavioral Therapy; CBT; Hypnosis
MeSH Terms: conditions — Breast Neoplasms; Affective Symptoms; Pathophobia; Emotional Regulation | interventions — Hypnosis

STUDY DESIGN:
Intervention Model Description: This is a two-armed, randomized, waiting-list controlled trial. Patients who agree to participate in the study will be randomly assigned to two groups: 1) the experimental group (EG) where six patients will receive one individual pre-group session and 8 sessions of group intervention combining cognitive-behavioral therapy and hypnosis; and 2) the waiting-list control group (CG) where six patients will receive the same intervention 4 months later. Patients will be assessed at three time points: 1) at baseline (T1), 2) 4 months later (T2), that means just after the intervention for the experimental group (EG) and just before the intervention for the control group (CG), and 3) 4 months later (T3), that means 4 months after the T2 for the experimental group and just after the intervention for the control group (CG).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Other): Patients include in the experimental group (EG) will receive one individual pre-group session and 8 sessions of group intervention combining cognitive-behavioral therapy and hypnosis after the first assessment (T1) (i.e., before the second assessment taking place 4 months later (T2)). They will resort to usual care only after the second assessment (T2) (i.e., before the third assessment taking place 4 months later (T3)).
  Interventions: Behavioral: Cognitive-Behavioral Group Therapy and Hypnosis
- Waiting-List Control Group (Other): Patients include in the waiting-list control group (CG) will resort to usual care only after the first assessment (T1) (i.e., before the second assessment taking place 4 months later (T2)). They will receive one individual pre-group session and 8 sessions of group intervention combining cognitive-behavioral therapy and hypnosis after the second assessment (T2) (i.e., before the third assessment taking place 4 months later (T3)).
  Interventions: Behavioral: Cognitive-Behavioral Group Therapy and Hypnosis

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Group Therapy and Hypnosis — The intervention consists in a pre-group interview and eight 2,5 h-session extended over 4 months. The intervention is based on cognitive-behavioral group therapy and hypnosis. To promote use of hypnosis at home, patients will receive audiorecordings of the hypnosis exercises. Starting immediately after the pre-group interview, the group will receive 3 app prompts a day promoting self-awareness and modulation of internal states, orientation of attention toward positive stimuli and inviting them to increase physical activity. Patients will be given a patient manual to promote an active approach to changes.
  Arms: Experimental Group
Behavioral: Cognitive-Behavioral Group Therapy and Hypnosis — The intervention consists in a pre-group interview and eight 2,5 h-session extended over 4 months. The intervention is based on cognitive-behavioral group therapy and hypnosis. To promote use of hypnosis at home, patients will receive audiorecordings of the hypnosis exercises. Starting immediately after the pre-group interview, the group will receive 3 app prompts a day promoting self-awareness and modulation of internal states, orientation of attention toward positive stimuli and inviting them to increase physical activity. Patients will be given a patient manual to promote an active approach to changes.
  Arms: Waiting-List Control Group

SUMMARY:
The end of treatment marks the beginning of a challenging period for breast cancer patients. While this period often provokes a sense of relief, it can also be a source of apprehension and vulnerability regarding the future. Patients may be brought to feel contradictory thoughts and emotions impacting their quality of life such as anxiety linked to uncertainty and fear of cancer recurrence. In order to accompany breast cancer patients during this transition period and to address these emotional difficulties, the Institut Jules Bordet has launched an 8-session psychological multi-component group intervention. Its objective is to bring patients tools and competencies (e.g., hypnosis, treatment of intrusive thoughts, learning to cope with uncertainty, attention reorientation toward positive thoughts) to promote emotion management and well-being.

DETAILED DESCRIPTION:
1. Introduction

   At the end of treatment, breast cancer patients are confronted with the short- and long-term physical (e.g., fatigue, pain, hot flashes) and psychological (e.g., anxiety, fear of recurrence, depressive symptoms) consequences of cancer diagnosis and treatment (Costanzo et al., 2007 ; Stanton et al., 2005). Emotion dysregulation (e.g., anxiety, fear of recurrence (Devine & Westlake,1995), depressive symptoms (Stanton, 2006)) is, with fatigue (Jacobsen & Jim, 2008) and cognitive dysfunctions (Duijts et al., 2011), one of the three most common complaints. Nevertheless, few psychological interventions have focused on this period (Jacobsen & Jim, 2008 ; Stanton et al., 2005 ; Stanton, 2006) and no intervention has specifically addressed emotion regulation of breast cancer survivors (Devine & Westlake, 1995 ; Duijts et al., 2011 ; Sheard & Maguire, 1999).

   Little is known about the required components of psychological interventions designed to support patients facing these challenges. Meta-analyses (Naaman et al., 2009 ; Osborn, 2006 ; Sheard & Maguire, 1999) and one review (Traeger et al., 2012) have described various components of interventions used to address anxiety and depressive symptoms in cancer care, such as mindfulness (Lengacher et al., 2009 ; Würtzen et al., 2013), education (Björneklett et al., 2012 ; Dolbeault et al., 2009 ; Duijts et al., 2011 ; Fors et al., 2011 ; Osborn, 2006 ; Scheier et al., 2005), cognitive-behavioral therapy (Dolbeault et al., 2009 ; Duijts et al., 2012 ; Fors et al., 2011 ; Osborn, 2006 ; Savard et al., 2005 ; Savard et al., 2005), support groups (Björneklett et al., 2012 ; Fors et al., 2011 ; Montazeri et al., 2001), and relaxation training (Björneklett et al., 2012 ; Elsesser, Van Berkel & Sartory, 1994 ; Hidderley & Holt, 2004). These interventions taken individually presented moderate effect sizes (Naaman et al., 2009), suggesting the need to combine components.

   During the last four years, our team conducted a study designed to compare the benefits in terms of emotion regulation of a 15-session single-component group intervention (SGI) based only on support with those of a 15-session multi-component group intervention (MGI) combining support with cognitive-behavioral and hypnosis components. The cognitive-behavioral therapy (CBT) components were chosen because interventions using such components have shown larger effect sizes than interventions using other components in previous studies on the treatment of anxiety-related conditions (Chambless & Ollendick, 2001 ; Deacon & Abramowitz, 2004 ; Norton & Price, 2007 ; Osborn, 2006 ; Stewart & Chambless, 2009). The hypnosis component was chosen because some reviews have suggested that self-hypnosis training is a rapid, cost-effective, and safe alternative to medication for the treatment of such conditions. Moreover, a meta-analysis showed that the addition of hypnosis to cognitive-behavioral component enhances effect sizes of interventions (Kirsch, Montgomery & Sapirstein, 1995) . Results of this study have shown the acceptability of such an intervention after active treatment (Merckaert et al., 2015). They have also indicated that an MGI combining support with CBT and hypnosis is clinically useful for patients with breast cancer after radiotherapy. Our results confirm the need to design specific interventions targeting anxiety regulation, fear of recurrence, and depressive symptoms. They also underline the necessity of intensifying interventions through including other components (e.g., emotion regulation, repetitive exposures to fear, treatment of intrusive thoughts, attention reorientation).
2. Objectives of the study

   The primary aims of this study are to evaluate in a randomized controlled trial (RCT) the efficacy of an 8-session multi-component group intervention extended over 4 months in promoting emotion regulation (in an emotion regulation task and in everyday life) and patient emotional well-being compared with a waiting-list control group. The secondary aims are to evaluate patients' satisfaction with the program, hypnosis/relaxation practice in everyday life, mental adjustment, and changes in patients' level of attentional bias toward cancer threat and physical activity.
3. Participants

   Patients who have been treated for a non-metastatic breast cancer will be approached at the end of active cancer treatment (i.e., surgery, chemotherapy, and radiotherapy) in order to be screened for emotion dysregulation. Patients experiencing moderate to high emotion dysregulation (one to four scores = or > 4 on a 11-point Likert adapted Edmonton symptoms evaluation scale assessing anxiety, fear of recurrence, depression, and intrusive thoughts) will be offered the intervention.
4. Intervention

4.1. Theoretical framework

This is a multi-component group intervention integrating an emotion regulation and an exposure to fear component.

4.1.1. The emotion regulation component builds upon the Adaptive Coping with Emotions Model which was developed to provide a conceptualization of adaptive emotion regulation. It aims to help patients to better identify their physical, emotional and behavioral responses to their positive and negative emotions in order to be able to better regulate or acknowledge those emotions. This component integrates a self-regulation component. The self-regulation component relies on a phone app-based coaching intervention aiming at promoting changes in patients' ability to regulate their emotions in their everyday life. It aims at promoting patients' self-awareness of their internal states, orientating their attention consciously toward positive stimuli and at developing physical activity. Hypnosis is used as hetero-hypnosis in each session and aims at deepening the development of patients' emotion regulation skills. Recordings of the exercises done in session are transmitted to the patients in order to promote use of the technique at home. Helping patients develop autohypnosis skills is important as it may allow them to better regulate their emotions in everyday life.

4.1.2. The exposure to fear component aims at helping patients deal with their fear of death. Just as anxiety is a normal emotion, anxiety concerning death is also a normal experience. The modest level of death anxiety that most people experience in everyday life may increase dramatically when one experiences a period of health problems, illness, or death of someone close (Kastenbaum, 2000). This part of the intervention will be based on worry exposure. This part of the intervention targets cancer-related worry and is based on Borkovec's avoidance theory of worry (Borkovec et al., 1998). Worry is a predominantly cognitive-verbal activity that inhibits full emotional processing. As a result, disturbing emotional meanings of potentially dangerous and anxiously anticipated events cannot be fully tested or altered, making the repetitive processing of the feared stimuli probable (Foa & Kozak, 1986). Given that cancer-recurrence related-worry is typically characterized by the focus on one hypothetical future event, it follows that exposure with imagined stimuli could be a crucial component of the treatment of fear of recurrence. The intervention will be based on two exercises. In the first, patients will be accompanied through a hypnosis based exposure to a major trigger of fear of recurrence that is the anticipation of the cancer check-up. This exercise is designed to help patients experience the emotions which may arise in this context while being guided through their resolution and regulation. The second exercise aims at helping them overcome their fear of recurrence through discussing their worst-case scenario in the group. The scenario are then discussed in order to highlight which part of them could be modified because it is unrealistic or because patients have more resources than they anticipate.

4.2. Study design and assessment schedule

This is a two-armed, randomized, waiting-list controlled trial. Patients who agree to participate will be randomly assigned to two groups: 1) the experimental group (EG) where six patients will receive one individual pre-group session and 8 sessions of group intervention combining cognitive-behavioral therapy and hypnosis; and 2) the waiting-list control group (CG) where six patients will receive the same intervention 4 months later. Patients will be assessed at three time points: 1) at baseline (T1), 2) 4 months later (T2), that means just after the intervention for the experimental group (EG) and just before the intervention for the control group (CG), and 3) 4 months later (T3), that means 4 months after the T2 for the experimental group and just after the intervention for the control group (CG).

4.2.1. Pre-assessment screening

Before inclusion in the study, during the last weeks of treatment (T0), approached patients will complete a socio-demographic questionnaire, a screening of life habits and difficulties questionnaire, an adapted Edmonton symptom evaluation scale (Chang, Hwang & Feuerman, 2000) (assessing pain, fatigue, sleep disturbances, fatigue, difficulty concentrating, memory loss, feeling of malaise, hot flashes, depression, anxiety, fear of recurrence, and worry), the Hospital anxiety and depression scale (HADS) (Zigmond & Snaith, 1983), and the Fear of Cancer Recurrence Inventory Severity sub-scale (Simard & Savard, 2009). Patients will report medical information about their disease, previous and current treatment and prognosis. This screening allows checking for inclusion and exclusion criteria and comparing patients who accept and refuse the intervention.

4.2.2. Assessment procedure

Each assessment procedure (i.e., T1, T2, T3) includes three parts: an emotion regulation task, an ecological momentary assessment and an attentional bias task. Two months after T1 and T2, the experimental (EG) and control (CG) groups will be contacted once by phone to complete a phone-based questionnaire to assess their usual care use.

4.2.2.1. Emotion regulation task

This assessment procedure has been used in a previous project and provides a dynamic picture of patients' emotion regulation. Each assessment session will first involve completion of questionnaires and two emotion regulation exercises: (1) 4 min exposure to anxiety triggers through completion of the Mental Adjustment to Cancer Scale (Watson et al., 1988), followed by a 12-min self-relaxation exercise in which patients will be asked to relax by using their own strategies; and (2) 4 min exposure to anxiety triggers through completion of the Impact of Cancer Questionnaire (Zebrack et al., 2006), followed by a 12-min guided hypnosis exercise in which patients will be asked to listen to an audio recording of a hypnotic induction script. The subtasks will be separated by a period of questionnaires completion. Patients' emotion regulation will be measured physiologically (heart rate measurement) and psychologically (anxiety, sadness, fear of recurrence and energy state-levels).

4.2.2.2. Ecological momentary assessment (EMA)

Patients' emotion regulation in their everyday life will be assessed during 9 days through an ecological momentary assessment (EMA) procedure. Firstly, patients will be asked 5 times a day to select on a list of 20 emotions the 2 or 3 that they were experiencing during the minutes before they saw the notification. For each emotion experienced, they will have to report its intensity on a 10-point Likert scale ranging from 1 to 10. They will have to report to what extent they have felt able to control those emotions and have felt submerged by those emotions. They will report whether during those minutes they had been thinking about something other than what they were currently doing. They will have to answer with one of four options: no; yes, something pleasant; yes, something neutral; or yes, something unpleasant (Killingsworth & Gilbert, 2010). Finally, they will be asked their level of fatigue and energy. Prompts will be sent randomly from 9 AM to 7,5 PM through the use of the software from http://www.lifedatacorp.com/. Secondly, each evening for 9 consecutive days, patients will have to indicate on the same list of 20 emotions (10 positive and 10 negative emotions), the extent to which they have felt each of the 20 emotions in the past 24 hours and their level of fatigue, from 0 (not at all) to 4 (extremely) (Fredrickson et al., 2003). In order to insure confidentiality, subjects will be provided with an iPod Touch. The two first days of data collection will be used as a training for participants and only their responses on the 7 following days will be taken into consideration. Thirdly, patients will be provided with an armband to continuously record during those 9 days, their heart rate levels, physical activity levels (pedometer and accelerometer) and sleep patterns (Garmin vívoactive HR).

4.2.2.3. Attentional bias task

Patients will complete an attentional bias computer task assessing attentional orientation toward emotional information. An adaptive function of biased attentional orientation toward negative information is to facilitate detection of danger in the environment and to help the organism respond effectively to threatening situations (Bar-Haim et al., 2007). When anxiety symptoms become excessive, biased attentional orientation toward negative information may have detrimental effects on patients' cognitive (e.g., intrusive thoughts, misinterpretation), behavioral (e.g., body screening, future planning difficulties), emotional (e.g., negative affects, panic attacks), and physiological status (e.g., physiological stress activation), and may play a prominent role in the etiology and maintenance of anxiety disorders (Bar-Haim et al., 2007). Computer tasks have been used to study the threat-related attentional bias in anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Experiencing moderate to high emotion dysregulation (one to four scores = or > 4 on a 11-point Likert adapted Edmonton symptoms evaluation scale assessing anxiety, fear of recurrence, depression, and intrusive thoughts)
* Non-metastatic breast cancer
* Post chimiotherapy, radiotherapy, surgery treatment
* Age > 18 years
* Completing a written informed consent

Exclusion Criteria:

* Male
* Non-fluency in French
* Severe cognitive impairment
* Severe and/or acute psychiatric disorder.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Change in Patients' Subjective Emotion Regulation through six 10-cm visual analog scales assessing anxiety, sadness, fear of cancer recurrence, physical fatigue, psychological fatigue, and energy state-levels | Change from T1 (baseline) Patients' Subjective Emotion Regulation at T2 (4 months after T1) and maintenance at T3 (4 months after T2) for the EG; Change from T2 Patients' Subjective Emotion Regulation at T3 (4 months after T2) for the CG
  Change in patients' subjective emotion regulation will be examined using the Emotion Regulation Task. Patients are asked to self-report their anxiety, sadness, fear of cancer recurrence, physical fatigue, psychological fatigue, and energy state-levels just after both exposures to anxiety triggers (the Mental Adjustment to Cancer Scale (MAC)) and the Impact of Cancer questionnaire Version 2 (IOCv2)) and regulation exercises (self-relaxation and induced relaxation) using six 10-cm visual analog scales (VAS; with the extreme left defined as "not at all" and the extreme right defined as "extremely"). VAS are used because such scales have been shown to be appropriate and adequate for the assessment of emotional states (Davey et al., 2007; Wewers & Lowe, 1990).
Change in Patients' Objective Emotion Regulation through an ambulatory digital Holter recording heart rate (beats per minute) | Change from T1 (baseline) Patients' Objective Emotion Regulation at T2 (4 months after T1) and maintenance at T3 (4 monts after T2) for the EG; Change from T2 Patients' Objective Emotion Regulation at T3 (4 monts after T2) for the CG
  Change in patients' objective emotion regulation will be examined using the Emotion Regulation Task. Heart rate (beats per minute) is measured throughout the Emotion Regulation Task using an ambulatory digital Holter recorder.
Change in Patients' Emotion Regulation in their Everyday Life through an ecological momentary assessment | Change from T1 (baseline) Emotion Regulation in their Everyday Life at T2 (4 months after T1) and maintenance at T3 (4 months after T2) for the EG; Change from T2 Emotion Regulation in their Everyday Life at T3 (4 months after T2) for the CG
  Change in patients' emotion regulation in their everyday life will be assessed through an ecological momentary assessment (EMA) procedure during 7 days. The EMA procedure will allow to observe the evolution of the ratio between positive and negative emotions in patients' everyday life (Fredrickson & Losada, 2005).
Change in Patients' Anxiety State through the Hospital Anxiety Depression Scale (HADS) - anxiety subscale and the Penn State Worry Questionnaire (PSWQ) | Change from T1 (baseline) Anxiety State at T2 (4 months after T1) and maintenance at T3 (4 months after T2) for the EG; Change from T2 Anxiety State at T3 (4 months after T2) for the CG
  Change in patients' emotional state will be assessed in terms of anxiety:
  Anxiety is assessed by the Hospital Anxiety Depression Scale (HADS) - anxiety 7-item ordinal self-report subscale (Duijts et al., 2012 ; Naaman et al., 2009). Each item is scored from 0 to 3. The subscale score ranges from 0 to 21. A subscale score from 0 to 7 is considered as normal, from 8 to 10 as an adaptation disorder, and from 11 to 21 as a mood disorder.
  Anxiety is also assessed by the 16-item ordinal self-report Penn State Worry Questionnaire (PSWQ; Meyer et al., 1990). Each item is scored from 1 ("not at all typical of me") to 5 ("very typical of me"). The total scale score ranges from 16 to 80, with higher scores reflecting greater levels of pathological worry.
Change in Patients' Depression State through the Hospital Anxiety Depression Scale (HADS) | Change from T1 (baseline) Depression State at T2 (4 months after T1) and maintenance at T3 (4 months after T2) for the EG; Change from T2 Depression State at T3 (4 months after T2) for the CG
  Change in patients' emotional state will be assessed in terms of depression:
  Depression is assessed by the Hospital Anxiety Depression Scale - depression 7-item ordinal self-report subscale (Duijts et al., 2012 ; Naaman et al., 2009). Each item is scored from 0 to 3. The subscale score ranges from 0 to 21. A subscale score from 0 to 7 is considered as normal, from 8 to 10 as an adaptation disorder, and from 11 to 21 as a mood disorder.
Change in Patients' Fear of Cancer Recurrence State through the Fear of Cancer Recurrence Inventory (FCRI) | Change from T1 (baseline) Fear of Cancer Recurrence State at T2 (4 months after T1) and maintenance at T3 (4 months after T2) for the EG; Change from T2 Fear of Cancer Recurrence State at T3 (4 months after T2) for the CG
  Change in patients' emotional state will be assessed in terms of fear of cancer recurrence: Fear of cancer recurrence is assessed by the Fear of Cancer Recurrence Inventory (FCRI). It is a 42-item 5-point ordinal self-report scale including seven subscales: triggers, severity, psychological distress, coping strategies, functioning impairments, insight, and reassurance (Simard & Savard, 2009). A higher score indicates higher levels of fear of cancer recurrence.

SECONDARY OUTCOMES:
Change in an adapted Emotion Symptom Assessment Scale (ESAS) | Change from T1 (baseline) ESAS at T2 (4 months after T1) and maintenance at T3 (4 months after T2) for the EG; Change from T2 ESAS at T3 (4 months after T2) for the CG
  Patients will complete a self-report adapted Emotion Symptom Assessment Scale (ESAS) assessing from 0 to 10 their usual emotional and symptomatic states (i.e., pain, physical fatigue, psychological fatigue, sleeping difficulties, memory disorder, concentration disorder, feeling of discomfort, hot flushes, depression, anxiety, fear of cancer recurrence, and ruminations).
Change in the Hospital Anxiety and Depression Scale (HADS) Questionnaire | Change from T1 (baseline) HADS at T2 (4 months after T1) and maintenance at T3 (4 months after T2) for the EG; Change from T2 HADS at T3 (4 months after T2) for the CG
  Patients will complete the Hospital Anxiety and Depression Scale (HADS) - anxiety and depression 14-item ordinal self-report subscales (Zigmond & Snaith, 1983). Each item is scored from 0 to 3. The total score ranges from 0 to 42. A total score from 0 to 12 is considered as normal, from 13 to 18 as an adaptation disorder, and from 19 to 42 as a mood disorder.
Change in the Fear of Cancer Recurrence Inventory (FCRI) Questionnaire | Change from T1 (baseline) FCRI at T2 (4 months after T1) and maintenance at T3 (4 months after T2) for the EG; Change from T2 FCRI at T3 (4 months after T2) for the CG
  Patients will complete the Fear of Cancer Recurrence Inventory (FCRI) (Simard & Savard, 2009). It is a 42-item 5-point ordinal self-report scale including seven subscales: triggers, severity, psychological distress, coping strategies, functioning impairments, insight, and reassurance (Simard & Savard, 2009). A higher score indicates higher levels of fear of cancer recurrence.
Change in the White Bear Suppression Inventory (WBSI) | Change from T1 (baseline) WBSI at T2 (4 months after T1) and maintenance at T3 (4 months after T2) for the EG; Change from T2 WBSI at T3 (4 months after T2) for the CG
  Patients will complete the White Bear Suppression Inventory (WBSI) (Schmidt et al., 2009 ; Wegner & Zanakos, 1994). The WBSI is a 15-item ordinal self-report measure of thought suppression. Each item is scored from 1 (strongly disagree) to 5 (strongly agree). Higher scores indicate greater tendencies to suppress thoughts.
Change in the Mental Adjustment to Cancer Scale (MAC) | Change from T1 (baseline) MAC at T2 (4 months after T1) and maintenance at T3 (4 months after T2) for the EG; Change from T2 MAC at T3 (4 months after T2) for the CG
  Patients will complete the Mental Adjustment to Cancer Scale (MAC) (Watson et al., 1988). The MAC is a 40-item ordinal self-report ordinal measure of five psychological dimensions of mental adjustment in cancer patients (fighting spirit, anxious preoccupation, helpless-hopelessness, fatalism, and avoidance). Each item is scored from 1 (definitely does not apply to me) to 4 (definitely applies to me).
Change in Penn State Worry Questionnaire (PSWQ) | Change from T1 (baseline) PSWQ at T2 (4 months after T1) and maintenance at T3 (4 months after T2) for the EG; Change from T2 PSWQ at T3 (4 months after T2) for the CG
  Patients will complete the 16-item ordinal self-report Penn State Worry Questionnaire (PSWQ; Meyer et al., 1990). Each item is scored from 1 ("not at all typical of me") to 5 ("very typical of me"). The total scale score ranges from 16 to 80, with higher scores reflecting greater levels of pathological worry.
Change in the Five Facet of Mindfulness Questionnaire (FFMQ) | Change from T1 (baseline) FFMQ at T2 (4 months after T1) and maintenance at T3 (4 months after T2) for the EG; Change from T2 FFMQ at T3 (4 months after T2) for the CG
  Patients will complete the Five Facet of Mindfulness Questionnaire (FFMQ) (Baer et al., 2008). The FFMQ is 39-item ordinal self-report measure of five facets of mindfulness: observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience. Each item is scored from 1 (never or very rarely true) to 5 (very often or always true), with higher scores indicating more mindfulness.
Change in the Metacognitions About Health Anxiety Questionnaire (MCQ-30) | Change from T1 (baseline) MCQ-30 at T2 (4 months after T1) and maintenance at T3 (4 months after T2) for the EG; Change from T2 MCQ-30 at T3 (4 months after T2) for the CG
  Patients will complete the Metacognitions About Health Anxiety Questionnaire (MCQ-30) (Wells & Cartwright-Hatton, 2004). The MCQ-30 is a 30-item self-report measure of metacognitive beliefs (beliefs about thinking). The MCQ-30 have five subscales: cognitive confidence, positive beliefs about worry, cognitive self-consciousness, negative beliefs about uncontrollability of thoughts and danger, and beliefs about the need to control thoughts. Each item is scored from 1 (do not agree) to 4 (agree very much). Subscale scores range from 6 to 24, and total scores range from 30 to 120, with higher scores indicating higher levels of unhelpful metacognitions.
Change in the Insomnia Severity Index (ISI) | Change from T1 (baseline) ISI at T2 (4 months after T1) and maintenance at T3 (4 months after T2) for the EG; Change from T2 ISI at T3 (4 months after T2) for the CG
  Patients will complete the Insomnia Severity Index (ISI) (Morin et al., 2011). The ISI is a brief 7-item self-report measure of insomnia. A total score from 0 to 7 is considered as no clinically significant insomnia, from 8 to 14 as a subthreshold insomnia, from 15 to 21 as a moderate clinical insomnia, and from 22 to 28 as a severe clinical insomnia.
Change in the Impact of Cancer Scale (IOCv2) | Change from T1 (baseline) IOCv2 at T2 (4 months after T1) and maintenance at T3 (4 months after T2) for the EG; Change from T2 IOCv2 at T3 (4 months after T2) for the CG
  Patients will complete the Impact of Cancer Scale (IOCv2) (Zebrack et al., 2006). The IOCv2 is a 37-item self-report measure of the quality of life of long-term cancer survivorship. The IOCv2 consists of two higher-order scales, a Positive Impact Scale and a Negative Impact Scale, each with four subscales: Altruism and empathy, health awareness, meaning of cancer, and positive self-evaluation subscales for the Positive Impact Scale, and appearance concerns, body change concerns, life interferences, and worry subscales for the Negative Impact Scale. The IOCv2 also have three additional subscales measuring employment and relationship impacts. Each item is scored from 1 (strongly disagree) to 5 (strongly agree). A higher score on a subscale/scale implies stronger endorsement of that content area.
Change in the Cognitive Emotion Regulation Questionnaire (CERQ) | Change from T1 (baseline) CERQ at T2 (4 months after T1) and maintenance at T3 (4 months after T2) for the EG; Change from T2 CERQ at T3 (4 months after T2) for the CG
  Patients will complete the Cognitive Emotion Regulation Questionnaire (CERQ) (Jermann et al., 2006). The CERQ is a 36-item self-report measure of cognitive emotion regulation strategies someone uses after having experienced negative events or situations. The CERQ distinguishes 9 cognitive coping strategie: Self-blame, acceptance, rumination, positive refocusing, refocus on planning, positive reappraisal, putting into perspective, catastrophizing, and other-blame. Each item is scored from 1 ((almost) never) to 5 (always). The higher the score on a subscale, the more the patient uses this cognitive coping strategy.
Change in the Multidimensional Fatigue Inventory (MFI-20) | Change from T1 (baseline) MFI-20 at T2 (4 months after T1) and maintenance at T3 (4 months after T2) for the EG; Change from T2 MFI-20 at T3 (4 months after T2) for the CG
  Patients will complete the Multidimensional Fatigue Inventory (MFI-20) (Smets et al., 1995). The MFI-20 is a 20-item self-report measure of fatigue which covers the five following dimensions: General fatigue, physical fatigue, mental fatigue, reduced motivation and reduced activity. Each item is scored from 1 (strongly disagree) to 5 (strongly agree). Higher scores indicating greater fatigue.
Change in a Life Event Questionnaire | Change from T1 (baseline) Life Event Questionnaire at T2 (4 months after T1) and maintenance at T3 (4 months after T2) for the EG; Change from T2 Life Event Questionnaire at T3 (4 months after T2) for the CG
  Patients will complete a life event questionnaire assessing hours of physical activity practice, hours of sleep, drugs use, cafeine, theine and alcohol intake, psychogical background, and health care use.
Change in Ecological Momentary Assessment through the use of a pedometer and a measure of cardio frequency (Garmin vívoactive® HR) | Change from T1 (baseline) Heart Rate, Physical Activiy and Sleep Patterns at T2 (4 months after T1) and maintenance at T3 (4 months after T2) for the EG; Change from T2 Ecological Momentary Assessment at T3 (4 months after T2) for the CG
  Patients are provided with an armband (Garmin vívoactive® HR) to continuously record during nine days (two days of test and seven days of assessment), their heart rate levels, physical activity levels (pedometer and accelerometer) and sleep patterns.
Change in Attentional Bias through a dot probe task | Change from T1 (baseline) Attentional Bias at T2 (4 months after T1) and maintenance at T3 (4 months after T2) for the EG; Change from T2 Attentional Bias at T3 (4 months after T2) for the CG
  The attentional dot probe computer task will provide a dynamic picture of patients' attentional orientation.

CONTACTS AND LOCATIONS:
Overall Officials: Darius Razavi, Prof, Principal Investigator — Université Libre de Bruxelles, Institut Jules Bordet; Isabelle Merckaert, Prof, Principal Investigator — Université Libre de Bruxelles, Institut Jules Bordet
Locations (1):
- Institut Jules Bordet, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Costanzo ES, Lutgendorf SK, Mattes ML, Trehan S, Robinson CB, Tewfik F, Roman SL. Adjusting to life after treatment: distress and quality of life following treatment for breast cancer. Br J Cancer. 2007 Dec 17;97(12):1625-31. doi: 10.1038/sj.bjc.6604091. Epub 2007 Nov 13. PMID 18000503
- [Background] Stanton AL, Ganz PA, Rowland JH, Meyerowitz BE, Krupnick JL, Sears SR. Promoting adjustment after treatment for cancer. Cancer. 2005 Dec 1;104(11 Suppl):2608-13. doi: 10.1002/cncr.21246. PMID 16247779
- [Background] Devine EC, Westlake SK. The effects of psychoeducational care provided to adults with cancer: meta-analysis of 116 studies. Oncol Nurs Forum. 1995 Oct;22(9):1369-81. PMID 8539178
- [Background] Stanton AL. Psychosocial concerns and interventions for cancer survivors. J Clin Oncol. 2006 Nov 10;24(32):5132-7. doi: 10.1200/JCO.2006.06.8775. PMID 17093275
- [Background] Jacobsen PB, Jim HS. Psychosocial interventions for anxiety and depression in adult cancer patients: achievements and challenges. CA Cancer J Clin. 2008 Jul-Aug;58(4):214-30. doi: 10.3322/CA.2008.0003. Epub 2008 Jun 16. PMID 18558664
- [Background] Duijts SF, Faber MM, Oldenburg HS, van Beurden M, Aaronson NK. Effectiveness of behavioral techniques and physical exercise on psychosocial functioning and health-related quality of life in breast cancer patients and survivors--a meta-analysis. Psychooncology. 2011 Feb;20(2):115-26. doi: 10.1002/pon.1728. PMID 20336645
- [Background] Sheard T, Maguire P. The effect of psychological interventions on anxiety and depression in cancer patients: results of two meta-analyses. Br J Cancer. 1999 Aug;80(11):1770-80. doi: 10.1038/sj.bjc.6690596. PMID 10468295
- [Background] Lang PJ, Davis M, Ohman A. Fear and anxiety: animal models and human cognitive psychophysiology. J Affect Disord. 2000 Dec;61(3):137-59. doi: 10.1016/s0165-0327(00)00343-8. PMID 11163418
- [Background] Stark DP, House A. Anxiety in cancer patients. Br J Cancer. 2000 Nov;83(10):1261-7. doi: 10.1054/bjoc.2000.1405. PMID 11044347
- [Background] Traeger L, Greer JA, Fernandez-Robles C, Temel JS, Pirl WF. Evidence-based treatment of anxiety in patients with cancer. J Clin Oncol. 2012 Apr 10;30(11):1197-205. doi: 10.1200/JCO.2011.39.5632. Epub 2012 Mar 12. PMID 22412135
- [Background] Bar-Haim Y, Lamy D, Pergamin L, Bakermans-Kranenburg MJ, van IJzendoorn MH. Threat-related attentional bias in anxious and nonanxious individuals: a meta-analytic study. Psychol Bull. 2007 Jan;133(1):1-24. doi: 10.1037/0033-2909.133.1.1. PMID 17201568
- [Background] Lebel S, Rosberger Z, Edgar L, Devins GM. Emotional distress impacts fear of the future among breast cancer survivors not the reverse. J Cancer Surviv. 2009 Jun;3(2):117-27. doi: 10.1007/s11764-009-0082-5. Epub 2009 Mar 26. PMID 19322661
- [Background] Llewellyn CD, Weinman J, McGurk M, Humphris G. Can we predict which head and neck cancer survivors develop fears of recurrence? J Psychosom Res. 2008 Dec;65(6):525-32. doi: 10.1016/j.jpsychores.2008.03.014. Epub 2008 Sep 24. PMID 19027440
- [Background] Baker F, Denniston M, Smith T, West MM. Adult cancer survivors: how are they faring? Cancer. 2005 Dec 1;104(11 Suppl):2565-76. doi: 10.1002/cncr.21488. PMID 16258929
- [Background] Armes J, Crowe M, Colbourne L, Morgan H, Murrells T, Oakley C, Palmer N, Ream E, Young A, Richardson A. Patients' supportive care needs beyond the end of cancer treatment: a prospective, longitudinal survey. J Clin Oncol. 2009 Dec 20;27(36):6172-9. doi: 10.1200/JCO.2009.22.5151. Epub 2009 Nov 2. PMID 19884548
- [Background] Harrison SE, Watson EK, Ward AM, Khan NF, Turner D, Adams E, Forman D, Roche MF, Rose PW. Primary health and supportive care needs of long-term cancer survivors: a questionnaire survey. J Clin Oncol. 2011 May 20;29(15):2091-8. doi: 10.1200/JCO.2010.32.5167. Epub 2011 Apr 25. PMID 21519023
- [Background] Sanson-Fisher R, Girgis A, Boyes A, Bonevski B, Burton L, Cook P. The unmet supportive care needs of patients with cancer. Supportive Care Review Group. Cancer. 2000 Jan 1;88(1):226-37. doi: 10.1002/(sici)1097-0142(20000101)88:13.3.co;2-g. PMID 10618627
- [Background] Hopwood P, Sumo G, Mills J, Haviland J, Bliss JM; START Trials Management Group. The course of anxiety and depression over 5 years of follow-up and risk factors in women with early breast cancer: results from the UK Standardisation of Radiotherapy Trials (START). Breast. 2010 Apr;19(2):84-91. doi: 10.1016/j.breast.2009.11.007. Epub 2009 Dec 29. PMID 20042336
- [Background] Lebel S, Rosberger Z, Edgar L, Devins GM. Comparison of four common stressors across the breast cancer trajectory. J Psychosom Res. 2007 Sep;63(3):225-32. doi: 10.1016/j.jpsychores.2007.02.002. Epub 2007 Aug 2. PMID 17719358
- [Background] Visser MR, Smets EM. Fatigue, depression and quality of life in cancer patients: how are they related? Support Care Cancer. 1998 Mar;6(2):101-8. doi: 10.1007/s005200050142. PMID 9540167
- [Background] DiMatteo MR, Lepper HS, Croghan TW. Depression is a risk factor for noncompliance with medical treatment: meta-analysis of the effects of anxiety and depression on patient adherence. Arch Intern Med. 2000 Jul 24;160(14):2101-7. doi: 10.1001/archinte.160.14.2101. PMID 10904452
- [Background] Falagas ME, Zarkadoulia EA, Ioannidou EN, Peppas G, Christodoulou C, Rafailidis PI. The effect of psychosocial factors on breast cancer outcome: a systematic review. Breast Cancer Res. 2007;9(4):R44. doi: 10.1186/bcr1744. PMID 17640330
- [Background] Bjorneklett HG, Lindemalm C, Rosenblad A, Ojutkangas ML, Letocha H, Strang P, Bergkvist L. A randomised controlled trial of support group intervention after breast cancer treatment: results on anxiety and depression. Acta Oncol. 2012 Feb;51(2):198-207. doi: 10.3109/0284186X.2011.610352. Epub 2011 Sep 19. PMID 21923569
- [Background] Naaman SC, Radwan K, Fergusson D, Johnson S. Status of psychological trials in breast cancer patients: a report of three meta-analyses. Psychiatry. 2009 Spring;72(1):50-69. doi: 10.1521/psyc.2009.72.1.50. PMID 19366294
- [Background] Osborn RL, Demoncada AC, Feuerstein M. Psychosocial interventions for depression, anxiety, and quality of life in cancer survivors: meta-analyses. Int J Psychiatry Med. 2006;36(1):13-34. doi: 10.2190/EUFN-RV1K-Y3TR-FK0L. PMID 16927576
- [Background] Lengacher CA, Johnson-Mallard V, Post-White J, Moscoso MS, Jacobsen PB, Klein TW, Widen RH, Fitzgerald SG, Shelton MM, Barta M, Goodman M, Cox CE, Kip KE. Randomized controlled trial of mindfulness-based stress reduction (MBSR) for survivors of breast cancer. Psychooncology. 2009 Dec;18(12):1261-72. doi: 10.1002/pon.1529. PMID 19235193
- [Background] Wurtzen H, Dalton SO, Elsass P, Sumbundu AD, Steding-Jensen M, Karlsen RV, Andersen KK, Flyger HL, Pedersen AE, Johansen C. Mindfulness significantly reduces self-reported levels of anxiety and depression: results of a randomised controlled trial among 336 Danish women treated for stage I-III breast cancer. Eur J Cancer. 2013 Apr;49(6):1365-73. doi: 10.1016/j.ejca.2012.10.030. Epub 2012 Dec 19. PMID 23265707
- [Background] Dolbeault S, Cayrou S, Bredart A, Viala AL, Desclaux B, Saltel P, Gauvain-Piquard A, Hardy P, Dickes P. The effectiveness of a psycho-educational group after early-stage breast cancer treatment: results of a randomized French study. Psychooncology. 2009 Jun;18(6):647-56. doi: 10.1002/pon.1440. PMID 19039808
- [Background] Scheier MF, Helgeson VS, Schulz R, Colvin S, Berga S, Bridges MW, Knapp J, Gerszten K, Pappert WS. Interventions to enhance physical and psychological functioning among younger women who are ending nonhormonal adjuvant treatment for early-stage breast cancer. J Clin Oncol. 2005 Jul 1;23(19):4298-311. doi: 10.1200/JCO.2005.05.362. PMID 15994143
- [Background] Fors EA, Bertheussen GF, Thune I, Juvet LK, Elvsaas IK, Oldervoll L, Anker G, Falkmer U, Lundgren S, Leivseth G. Psychosocial interventions as part of breast cancer rehabilitation programs? Results from a systematic review. Psychooncology. 2011 Sep;20(9):909-18. doi: 10.1002/pon.1844. Epub 2010 Sep 6. PMID 20821803
- [Background] Duijts SF, van Beurden M, Oldenburg HS, Hunter MS, Kieffer JM, Stuiver MM, Gerritsma MA, Menke-Pluymers MB, Plaisier PW, Rijna H, Lopes Cardozo AM, Timmers G, van der Meij S, van der Veen H, Bijker N, de Widt-Levert LM, Geenen MM, Heuff G, van Dulken EJ, Boven E, Aaronson NK. Efficacy of cognitive behavioral therapy and physical exercise in alleviating treatment-induced menopausal symptoms in patients with breast cancer: results of a randomized, controlled, multicenter trial. J Clin Oncol. 2012 Nov 20;30(33):4124-33. doi: 10.1200/JCO.2012.41.8525. Epub 2012 Oct 8. PMID 23045575
- [Background] Savard J, Simard S, Ivers H, Morin CM. Randomized study on the efficacy of cognitive-behavioral therapy for insomnia secondary to breast cancer, part I: Sleep and psychological effects. J Clin Oncol. 2005 Sep 1;23(25):6083-96. doi: 10.1200/JCO.2005.09.548. PMID 16135475
- [Background] Savard J, Simard S, Ivers H, Morin CM. Randomized study on the efficacy of cognitive-behavioral therapy for insomnia secondary to breast cancer, part II: Immunologic effects. J Clin Oncol. 2005 Sep 1;23(25):6097-106. doi: 10.1200/JCO.2005.12.513. PMID 16135476
- [Background] Montazeri A, Jarvandi S, Haghighat S, Vahdani M, Sajadian A, Ebrahimi M, Haji-Mahmoodi M. Anxiety and depression in breast cancer patients before and after participation in a cancer support group. Patient Educ Couns. 2001 Dec 1;45(3):195-8. doi: 10.1016/s0738-3991(01)00121-5. PMID 11722855
- [Background] Elsesser, K., Van Berkel, M., & Sartory, G. (1994). The effects of anxiety management training on psychological variables and immune parameters in cancer patients. Behavioural and Cognitive Psychotherapy, 22, 13-23.
- [Background] Hidderley M, Holt M. A pilot randomized trial assessing the effects of autogenic training in early stage cancer patients in relation to psychological status and immune system responses. Eur J Oncol Nurs. 2004 Mar;8(1):61-5. doi: 10.1016/j.ejon.2003.09.003. PMID 15003745
- [Background] Humphris G, Ozakinci G. The AFTER intervention: a structured psychological approach to reduce fears of recurrence in patients with head and neck cancer. Br J Health Psychol. 2008 May;13(Pt 2):223-30. doi: 10.1348/135910708X283751. PMID 18492319
- [Background] Lebel S, Maheu C, Lefebvre M, Secord S, Courbasson C, Singh M, Jolicoeur L, Benea A, Harris C, Fung MF, Rosberger Z, Catton P. Addressing fear of cancer recurrence among women with cancer: a feasibility and preliminary outcome study. J Cancer Surviv. 2014 Sep;8(3):485-96. doi: 10.1007/s11764-014-0357-3. Epub 2014 Apr 23. PMID 24756313
- [Background] Mishel MH, Germino BB, Gil KM, Belyea M, Laney IC, Stewart J, Porter L, Clayton M. Benefits from an uncertainty management intervention for African-American and Caucasian older long-term breast cancer survivors. Psychooncology. 2005 Nov;14(11):962-78. doi: 10.1002/pon.909. PMID 15712339
- [Background] Simard S, Thewes B, Humphris G, Dixon M, Hayden C, Mireskandari S, Ozakinci G. Fear of cancer recurrence in adult cancer survivors: a systematic review of quantitative studies. J Cancer Surviv. 2013 Sep;7(3):300-22. doi: 10.1007/s11764-013-0272-z. Epub 2013 Mar 10. PMID 23475398
- [Background] Herschbach P, Book K, Dinkel A, Berg P, Waadt S, Duran G, Engst-Hastreiter U, Henrich G. Evaluation of two group therapies to reduce fear of progression in cancer patients. Support Care Cancer. 2010 Apr;18(4):471-9. doi: 10.1007/s00520-009-0696-1. Epub 2009 Oct 29. PMID 19865833
- [Background] Chambless DL, Ollendick TH. Empirically supported psychological interventions: controversies and evidence. Annu Rev Psychol. 2001;52:685-716. doi: 10.1146/annurev.psych.52.1.685. PMID 11148322
- [Background] Deacon BJ, Abramowitz JS. Cognitive and behavioral treatments for anxiety disorders: a review of meta-analytic findings. J Clin Psychol. 2004 Apr;60(4):429-41. doi: 10.1002/jclp.10255. PMID 15022272
- [Background] Norton PJ, Price EC. A meta-analytic review of adult cognitive-behavioral treatment outcome across the anxiety disorders. J Nerv Ment Dis. 2007 Jun;195(6):521-31. doi: 10.1097/01.nmd.0000253843.70149.9a. PMID 17568301
- [Background] Stewart RE, Chambless DL. Cognitive-behavioral therapy for adult anxiety disorders in clinical practice: a meta-analysis of effectiveness studies. J Consult Clin Psychol. 2009 Aug;77(4):595-606. doi: 10.1037/a0016032. PMID 19634954
- [Background] Hammond DC. Hypnosis in the treatment of anxiety- and stress-related disorders. Expert Rev Neurother. 2010 Feb;10(2):263-73. doi: 10.1586/ern.09.140. PMID 20136382
- [Background] Kirsch I, Montgomery G, Sapirstein G. Hypnosis as an adjunct to cognitive-behavioral psychotherapy: a meta-analysis. J Consult Clin Psychol. 1995 Apr;63(2):214-20. doi: 10.1037//0022-006x.63.2.214. PMID 7751482
- [Background] Merckaert I, Lewis F, Delevallez F, Herman S, Caillier M, Delvaux N, Libert Y, Lienard A, Nogaret JM, Ogez D, Scalliet P, Slachmuylder JL, Van Houtte P, Razavi D. Improving anxiety regulation in patients with breast cancer at the beginning of the survivorship period: a randomized clinical trial comparing the benefits of single-component and multiple-component group interventions. Psychooncology. 2017 Aug;26(8):1147-1154. doi: 10.1002/pon.4294. Epub 2016 Nov 7. PMID 27718533
- [Background] Berking, M., & Schwarz, J. (2013). Affect regulation training. Handbook of Emotion Regulation. New York: Guilford.
- [Background] Kastenbaum, R. (2000). The psychology of death (3rd ed.). New York: Springer.
- [Background] Borkovec, T.D., et al. (1998). Worry: a cognitive phenomenon intimately linked to affective, physiological, and interpersonal behavioral processes. Cognitive Therapy and Research, 22(6), 561-576.
- [Background] Foa EB, Kozak MJ. Emotional processing of fear: exposure to corrective information. Psychol Bull. 1986 Jan;99(1):20-35. No abstract available. PMID 2871574
- [Background] Merckaert, I., et al. (2016). Emotion regulation at the beginning of the survivorship period for breast cancer: Comparing the impact of an 8-session to a 15-session multicomponent group intervention, submitted abstract. Psychooncology.
- [Background] Chang VT, Hwang SS, Feuerman M. Validation of the Edmonton Symptom Assessment Scale. Cancer. 2000 May 1;88(9):2164-71. doi: 10.1002/(sici)1097-0142(20000501)88:93.0.co;2-5. PMID 10813730
- [Background] Simard S, Savard J. Fear of Cancer Recurrence Inventory: development and initial validation of a multidimensional measure of fear of cancer recurrence. Support Care Cancer. 2009 Mar;17(3):241-51. doi: 10.1007/s00520-008-0444-y. Epub 2008 Apr 15. PMID 18414902
- [Background] Watson M, Greer S, Young J, Inayat Q, Burgess C, Robertson B. Development of a questionnaire measure of adjustment to cancer: the MAC scale. Psychol Med. 1988 Feb;18(1):203-9. doi: 10.1017/s0033291700002026. PMID 3363039
- [Background] Zebrack BJ, Ganz PA, Bernaards CA, Petersen L, Abraham L. Assessing the impact of cancer: development of a new instrument for long-term survivors. Psychooncology. 2006 May;15(5):407-21. doi: 10.1002/pon.963. PMID 16097041
- [Background] Killingsworth MA, Gilbert DT. A wandering mind is an unhappy mind. Science. 2010 Nov 12;330(6006):932. doi: 10.1126/science.1192439. PMID 21071660
- [Background] Fredrickson BL, Losada MF. Positive affect and the complex dynamics of human flourishing. Am Psychol. 2005 Oct;60(7):678-86. doi: 10.1037/0003-066X.60.7.678. PMID 16221001
- [Background] Zelenski, J. M., & Larsen, R. J. (2000). The Distribution of Basic Emotions in Everyday Life: A State and Trait Perspective from Experience Sampling Data. Journal of Research in Personality, 34(2), 178-197.
- [Background] Fredrickson BL. The role of positive emotions in positive psychology. The broaden-and-build theory of positive emotions. Am Psychol. 2001 Mar;56(3):218-26. doi: 10.1037//0003-066x.56.3.218. PMID 11315248
- [Background] Meyer TJ, Miller ML, Metzger RL, Borkovec TD. Development and validation of the Penn State Worry Questionnaire. Behav Res Ther. 1990;28(6):487-95. doi: 10.1016/0005-7967(90)90135-6. PMID 2076086
- [Background] Shiffman S, Stone AA, Hufford MR. Ecological momentary assessment. Annu Rev Clin Psychol. 2008;4:1-32. doi: 10.1146/annurev.clinpsy.3.022806.091415. PMID 18509902
- [Background] Davey HM, Barratt AL, Butow PN, Deeks JJ. A one-item question with a Likert or Visual Analog Scale adequately measured current anxiety. J Clin Epidemiol. 2007 Apr;60(4):356-60. doi: 10.1016/j.jclinepi.2006.07.015. Epub 2006 Dec 27. PMID 17346609
- [Background] Miller MD, Ferris DG. Measurement of subjective phenomena in primary care research: the Visual Analogue Scale. Fam Pract Res J. 1993 Mar;13(1):15-24. PMID 8484338
- [Background] Wewers ME, Lowe NK. A critical review of visual analogue scales in the measurement of clinical phenomena. Res Nurs Health. 1990 Aug;13(4):227-36. doi: 10.1002/nur.4770130405. PMID 2197679
- [Background] Friedman BH. An autonomic flexibility-neurovisceral integration model of anxiety and cardiac vagal tone. Biol Psychol. 2007 Feb;74(2):185-99. doi: 10.1016/j.biopsycho.2005.08.009. Epub 2006 Oct 27. PMID 17069959
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Schmidt RE, Gay P, Courvoisier D, Jermann F, Ceschi G, David M, Brinkmann K, Van der Linden M. Anatomy of the White Bear Suppression Inventory (WBSI): a review of previous findings and a new approach. J Pers Assess. 2009 Jul;91(4):323-30. doi: 10.1080/00223890902935738. PMID 20017061
- [Background] Baer RA, Smith GT, Lykins E, Button D, Krietemeyer J, Sauer S, Walsh E, Duggan D, Williams JM. Construct validity of the five facet mindfulness questionnaire in meditating and nonmeditating samples. Assessment. 2008 Sep;15(3):329-42. doi: 10.1177/1073191107313003. Epub 2008 Feb 29. PMID 18310597
- [Background] Wells A, Cartwright-Hatton S. A short form of the metacognitions questionnaire: properties of the MCQ-30. Behav Res Ther. 2004 Apr;42(4):385-96. doi: 10.1016/S0005-7967(03)00147-5. PMID 14998733
- [Background] Morin CM, Belleville G, Belanger L, Ivers H. The Insomnia Severity Index: psychometric indicators to detect insomnia cases and evaluate treatment response. Sleep. 2011 May 1;34(5):601-8. doi: 10.1093/sleep/34.5.601. PMID 21532953
- [Background] Jermann, F., et al. (2006). Cognitive Emotion Regulation Questionnaire (CERQ): Confirmatory Factor Analysis and Psychometric Properties of the French Translation. European Journal of Psychological Assessment, 22, 126-131.
- [Background] Smets EM, Garssen B, Bonke B, De Haes JC. The Multidimensional Fatigue Inventory (MFI) psychometric qualities of an instrument to assess fatigue. J Psychosom Res. 1995 Apr;39(3):315-25. doi: 10.1016/0022-3999(94)00125-o. PMID 7636775
- [Background] Killip S, Mahfoud Z, Pearce K. What is an intracluster correlation coefficient? Crucial concepts for primary care researchers. Ann Fam Med. 2004 May-Jun;2(3):204-8. doi: 10.1370/afm.141. PMID 15209195
- [Derived] Merckaert I, Waroquier P, Caillier M, Verkaeren O, Righes S, Lienard A, Libert Y, Kristanto P, Razavi D. Improving emotion regulation in breast cancer patients in the early survivorship period: Efficacy of a brief ecologically boosted group intervention. Psychooncology. 2023 Apr;32(4):597-609. doi: 10.1002/pon.6105. Epub 2023 Mar 8. PMID 36703250
- Available data/document: Study design — http://pdf.lu/YtWd
- Available data/document: List of questionnaires — http://pdf.lu/TJ4c
- Available data/document: Informed Consent Form — http://pdf.lu/dN2P
- Available data/document: Informed Consent Form — http://pdf.lu/07Xz